CLINICAL TRIAL: NCT00432146
Title: Positive Effect of Lugol's Solution on the Blood Flow and Microvessel Density of Thyroid Gland in the Patients With Graves' Disease
Brief Title: Effect of Lugol's Solution in the Patients With Graves' Disease
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Other Study IDs: 2005/117
Record Dates: First submitted 2007-02-05; First posted 2007-02-07 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2007-02

CONDITIONS: Graves Disease
Keywords: Graves' disease, Lugol's solution
MeSH Terms: conditions — Graves Disease | interventions — Lugol's solution

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: lugol's solution

SUMMARY:
Context: Although some of endocrine surgeons administer Lugol's solution to decrease thyroid gland vascularity, there is still no agreement on its effectiveness.

Objective: The aims of this clinical trial are to evaluate thyroid blood flow and microvessel density in the patients with Graves' disease according to the Lugol's solution treatment preoperatively.

Design: Retrospective clinical trial. Setting: A tertiary referral center. Method: Thirty-six patients were randomly assigned to preoperative medication with Lugol's solution. Patients in group 1 (n=17) received Lugol's solution for 10 days before surgical intervention, whereas patients in group 2 (n=19) didn't receive it.

Main Outcome Measures: Blood flow through the thyroid arteries of patients with Graves' disease was measured by color flow Doppler ultrasonography. The microvessel density (MVD) was assessed immunohistochemically and Western blot analysis using the level of expression of CD-34 in thyroid tissue. The thyroid gland's weight and blood loss were measured in all patients.

DETAILED DESCRIPTION:
Thirty-six patients were randomly assigned to preoperative medication with Lugol's solution. Patients in group 1 (n=17) received Lugol's solution for 10 days before surgical intervention, whereas patients in group 2 (n=19) didn't receive it. Blood flow through the thyroid arteries of patients with Graves' disease was measured by color flow Doppler ultrasonography. The microvessel density (MVD) was assessed immunohistochemically and Western blot analysis using the level of expression of CD-34 in thyroid tissue. The thyroid gland's weight and blood loss were measured in all patients.

ELIGIBILITY:
Inclusion Criteria:

* Graves disease

Exclusion Criteria:

* Anticoagulant usage,
* Previous thyroid operation,
* Refused to participate in this study.

Ages: 14 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36
Dates: Start 2005-09; Study Completion 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: yesim erbil, Study Director — Istanbul University